CLINICAL TRIAL: NCT03991052
Title: Controlled Mean Arterial Pressure of Brain Injury Patients Using an Novel Automated System for Vasopressor Administration : a Randomized Controlled Trial in Critically Ill Patients in the Intensive Care Unit
Brief Title: Controlled MAP in the Brain Injury Patient (COMAT Study)
Acronym: COMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP180501
Record Dates: First submitted 2019-05-24; First posted 2019-06-19 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: manual versus automated management of MAP
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV1000 monitor (Active Comparator): MAP management will be done as usual (adjustment by nurses) and fluid management will be managed using the EV1000 monitoring device with the automated decision support system
  Interventions: Device: Control group
- EV1000 monitor + closed-loop system (Experimental): Fluid management will be done using the automated decision support system and MAP will be adjusted by the automated closed-loop system for vasopressor administration
  Interventions: Device: EV1000 and closed-loop system

INTERVENTIONS:
Device: EV1000 and closed-loop system — This system will recommend when patients need fluid or not and adjust vasopressor administration automatically by the closed-loop system
  Arms: EV1000 monitor + closed-loop system
Device: Control group — This system will recommend when patients need fluid or not and nurses will adjust vasopressor administration as usual (standard of care)
  Arms: EV1000 monitor

SUMMARY:
The goal of this randomized controlled trial will be to show that the use of a novel automated system to guide vasopressor administration in brain injury patients will results in more time spent with a mean arterial pressure (MAP) within the predefined MAP (+/- 5 mmHg of the target MAP) compared to patients managed without any automated system (manually management)

DETAILED DESCRIPTION:
In brain injury patients, the maintenance of MAP within a very narrow range is desired to avoid complications related to hypoperfusion (undertreatment) or hypertension (over treatment). However, the MAP needed to reach can vary over time based on intracranial pressure. Additionally, it is well know that the nurses in the Intensive care unit managed multiple patients simultaneously and cannot dedicate 100% of his-her time to adjust drugs infusions. Using a novel automated system can overcome this issue and may lead to more time in MAP target (+/- 5mmHg) than the traditional management.

After initial rescuscitation of the patients, patients in both groups will have the same baseline maintenance fluid administration of 1-2 ml/kg/h of crystalloid solution and additionnal fluid boluses administered following the EV1000 monitoring device. The only difference will be the management of vasopressor titration (manual by nurses vs automated via a closed-loop system)

ELIGIBILITY:
Inclusion Criteria:

* severe brain injury patients (Glasgow score <9), intubated, ventilated and sedated.

Exclusion Criteria:

* Glasgow score > 8
* Bilateral mydriasis at the initial management (Ambulance and first hour of arrival)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) | 48 hours post-admission in the intensive care unit
  percentage of treatment time when MAP will be in the predefined range (+/- 5 mmHg of the target MAP)

SECONDARY OUTCOMES:
Percentage of case time spent in Hypotension | 48 hours post-admission in the intensive care unit
  percentage time spent with MAP below 5 mmHg of the predefined MAP
Percentage of case time spent Hypertension | 48 hours post-admission in the intensive care unit
  percentage time spent with MAP above 5 mmHg of the predefined MAP
Cerebral perfusion pressure | 48 hours post-admission in the intensive care unit
  Measure of Cerebral perfusion pressure during the treatment time (evolution of Cerebral perfusion pressure over time)
Intracranial pressure | 48 hours post-admission in the intensive care unit
  Measure of intracranial pressure during the treatment time (evolution over time)
Intracranial pressure Hypertension | 48 hours post-admission in the intensive care unit
  percentage of intracranial pressure over 20 mmHg during the treatment period
Fluid received | 48 hours post-admission in the intensive care unit
  comparison of amount of fluid received during the treatment period
Amount of vasopressor | 48 hours post-admission in the intensive care unit
  amount of vasopressor received during the treatment period
Length of stay in the intensive care unit | 30 days post-admission in the intensive care unit
  comparison of the length of stay in the intensive care unit between both groups.
mean arterial pressure (MAP) | 48 hours post-admission in the intensive care unit
  MAP over the treatment period
stroke volume | 48 hours post-admission in the intensive care unit
  stroke volume over the treatment period
cardiac index | 48 hours post-admission in the intensive care unit
  cardiac index over the treatment period. This will be the mean values over the procedure. Measurements recorded each 20 seconds and averaged for the procedure. The unit is l/min/m-2
Transcranial doppler | 48 hours post-admission in the intensive care unit
  measure of mean cerebral velocity of mean cerebral artery

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DURANTEAU, MD, PhD, Study Chair — Bicetre
Locations (1):
- Bicêtre hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No